CLINICAL TRIAL: NCT01784471
Title: A Pilot Study to Assess the Use of the Magic Foot in the Improvement of Subjective and Objective Parameters in Subjects With Foot Symptoms as a Result of Diabetes or Peripheral Vascular Disease.
Brief Title: Open-label Pilot Study to Assess the Use of Magic Foot™ in the Improvment of Parameters in Subject With Foot Symptoms
Acronym: MF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yaffa Golan, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MF-1
Record Dates: First submitted 2013-01-30; First posted 2013-02-05 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Peripheral Vascular Disease
Keywords: Foot Symptoms; Diabetes; Peripheral Vascular Disease; Magic Foot shoe
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magic foot shoe (Experimental): Magic Foot™ will be dispensed to all subjects. Shoes will be activated at the clinic for 30 minutes. Subjects will self-use and activate the shoes at home daily for 30 days.
  Interventions: Device: Magic Foot™

INTERVENTIONS:
Device: Magic Foot™ — Magic Foot™ is a shoe, providing massage together with acupressure or reflexology functions. The device is fully remotely operated and controlled.

SUMMARY:
This is a single-arm, single-center, open-label, pilot study . 30 subjects with foot symptoms attributable to diabetes or peripheral vascular disease will be screened . Subjects meeting inclusion criteria will sign informed consent and enrolled. All 30 subjects will be treated with the Magic Foot™.

If there is any significant improvement in ICG or foot symptoms as obtained from self evaluation questionnaire, a further 30 subjects will be enrolled.

DETAILED DESCRIPTION:
This is a single-arm, single-center, open-label, pilot study . 30 subjects with foot symptoms attributable to diabetes or peripheral vascular disease will be screened and enrolled. Subjects meeting inclusion criteria will sign informed consent. They will undergo a full examination including blood pressure measurement, heart rate and ECG.

A self evaluation questionnaire relating to foot and sleep disorder symptoms will be completed.

A baseline screening ICG will be performed to measure total peripheral resistance CO (Cardiac Output) and SV (Stroke Volume).

ABI will be performed. The investigational product will be used for 30 minutes and ICG will be repeated.

Each subject will be provided with a size appropriate pair of Magic Foot™ to use at home.

Magic Foot™ will be used for thirty minutes daily for 30 days. This will be done at rest in the evening prior to bedtime. A diary to report compliance will be provided to the subjects. The subject will provide the completed diary to the site staff at day 14 and day 30. Subjects will be reassessed at Day 14. Self evaluation questionnaire will be completed. Subjects will continue with daily use of Magic Foot™. Subject will be reassessed at day 30. ICG, ABI (Ankle Bracial Index) and a final self assessment questionnaire will be repeated at day 30.

At the end of the study the Magic Foot™ will remain with the subjects. In consultation with the treating physician a decision will be made whether to continue with treatment or not.

ELIGIBILITY:
Inclusion Criteria:

1. Subject over the age of 18 with Type 1 / Type 2 diabetes or with PVD (Peripheral vascular disease) or ABI < 0.9 with foot symptoms.
2. Subject able and willing to comply with the requirements of the protocol.
3. Subject able to understand and sign written informed consent to participate in the study.

One or more of the following foot symptoms:

* Pain at rest
* Pain on activity
* Nocturnal feet pain
* Burning sensations
* Loss of sensation
* Cold feet
* Recurrent ulcers , wounds , injuries - longtime to heal

Exclusion Criteria:

1. Active foot infection
2. Open ulcer in shoe area
3. Subjects with unstable or lifethreatening conditions
4. History of malignancy
5. Active Charcot arthropathy
6. Impaired cognitive function -unable to sign informed consent
7. History of drug or alcohol abuse
8. Subject currently enrolled or has not yet completed other investigational device or drug study or subject is receiving other investigational agents.
9. Other conditions based on Principle Investigators judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-03-14 (Actual)

PRIMARY OUTCOMES:
Changes in total peripheral resistance as assessed by impedance cardiography (ICG) from baseline to day 30 | From baseline to day 30.

CONTACTS AND LOCATIONS:
Overall Officials: Eliezer Klainman, M.D., Principal Investigator — Gefen Cardiac Health
Locations (1):
- Gefen Cardiac Health Center, Giv‘atayim, Israel